CLINICAL TRIAL: NCT01301469
Title: Prospective, Randomized, Double-blind, Controlled, Multicenter Study on the Efficacy and Safety of HES 130/0. 42 in a Balanced Electrolyte Solution vs a HES 130/0.4 in a Sodium Chloride Solution in Elective Surgery Patients
Brief Title: Comparison of HES 130 in Balanced and in Unbalanced Solution
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HC-G-H-0801
Record Dates: First submitted 2011-02-11; First posted 2011-02-23 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Decreased and Nonspecific Blood Pressure Disorders and Shock
MeSH Terms: conditions — Shock | interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 6% HES 130/0.42 in plasma adapted Ringer's solution (balanced solution)
  Interventions: Drug: 6% HES 130/0.42 in plasma adapted Ringer's solution
- 2 (Active Comparator): HES 130/0.4 in a saline solution
  Interventions: Drug: 6% HES 130/0.4 in a saline solution

INTERVENTIONS:
Drug: 6% HES 130/0.42 in plasma adapted Ringer's solution — 60 g/l hydroxyethyl starch 130 dissolved in plasma adapted Ringer's solution (balanced solution)
  Arms: 1
Drug: 6% HES 130/0.4 in a saline solution — 60 g/l Hydroxyethyl starch (HES) with a mean molecular weight of 130 kDalton which is dissolved in a saline solution
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of HES 130/0.42 in an electrolyte infusion in comparison to HES 130/0.4 in a sodium chloride infusion.

ELIGIBILITY:
Inclusion:

* Male or female (non pregnant) patients; between 18 and 70 years
* Elective non-cardiac surgery (except pancreatic or neurological surgery) with an estimated operation duration of 2 hours or longer
* General anesthesia
* Voluntary consent

Exclusion:

* Patients of ASA-class III or IV, Cardiac insufficiency NYHA classes III. IV
* BMI < 18 or > 29
* Patients with daily urine output < 1L
* Patients on hemodialysis
* Abnormal liver or renal function (i. e. above upper limit of normal range)
* Abnormal coagulation function (prothrombin time (PT) 3 seconds higher than normal or activated partial thromboplastin time (APTT) 10 seconds higher than normal)
* Hgb < 10g/dl or HCT < 30%
* Potassium, sodium or chloride above the upper limit of normal of the laboratory
* History of diabetes mellitus
* Known history of a mental or neurological disorder, such as epileptic seizures.
* History of hypertension and/or taking a beta-receptor blocker or history of atrial fibrillation
* Patients with known hypersensitivity and with contraindications to HES or any of the excipients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Maximum difference of the mean arterial blood pressure | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Buwei Yu, Prof. Dr., Principal Investigator — Ruijin Hospital
Locations (4):
- China (4):
  - 2 Hospitals, Beijing
  - Hospital, Guangzhou
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Hospital, Shanghai